CLINICAL TRIAL: NCT05409170
Title: Division of Plastic Surgery, Department of Surgery, Wan Fang Hospital, Taipei Medical University, Taipei, Taiwan
Brief Title: The Change of Clinical Features and Surgical Outcomes in Patients With Pressure Injury During the COVID-19 Pandemic: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Wen-Kuan Chiu, TMU-Joint Institutional Review Board, Taipei Medical University WanFang Hospital
Other Study IDs: WanFangW
Record Dates: First submitted 2022-06-07; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Pressure Injury; COVID-19
MeSH Terms: conditions — Pressure Ulcer; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pre-covid group: Each surgical procedure was considered an independent event. , the January 2016-December 2019 and January 2020-December 2021 intervals were defined as pre-COVID and COVID periods, respectively.
- covid group: Each surgical procedure was considered an independent event. , the January 2016-December 2019 and January 2020-December 2021 intervals were defined as pre-COVID and COVID periods, respectively.
  Interventions: Procedure: COVID

INTERVENTIONS:
Procedure: COVID — Each surgical procedure was considered an independent event. Moreover, the January 2016-December 2019 and January 2020-December 2021 intervals were defined as pre-COVID and COVID periods, respectively.
  Groups: covid group

SUMMARY:
The COVID-19 pandemic has considerably and negatively affected numerous lives and economies worldwide; specifically, it has led to delays in seeking medical treatment among many people [1-3]. Delaying or avoiding seeking medical advice can result in worsened symptoms, delayed evaluation, and treatment complications [4-7]. Moreover, the pandemic has significantly impacted health-care systems, leading to numerous issues including shortages of medical staff, beds, equipment, medicines, and isolation facilities. The concern of cross-contamination-where COVID-19 may spread within wards unknowingly-has also increased the emotional burden among health-care workers [8-10].

Pressure injury (PI) is a common health issue particularly among older people who have physical limitations or are bedridden. PI management often requires a long-term individualized plan. Failure to implement this strategy may influence the quality of life and may cause wound-related psychosocial issues (e.g., low self-esteem), increase health-care expenditures, and shorten survival among the patients [11]. Moreover, long-term PIs are prone to infection and bleeding, which may lead to sepsis or anemia [12-14].

The current study explored whether COVID-19 pandemic-related changes affected the characteristics and treatment outcomes of patients with PIs.

ELIGIBILITY:
Inclusion Criteria:

* all patients who received debridement or flap-reconstruction surgery for Pressure injury at Wan Fang Hospital from January 2016 to December 2021.

Exclusion Criteria:

* Patients who underwent debridement or flap-reconstruction surgery across the pre-COVID and COVID periods were excluded from the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the January 2016-December 2019 and January 2020-December 2021 intervals were defined as pre-COVID and COVID periods, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
flap surgery outcomes | from January 2016 to December 2021
  complete wound healing, major and minor complications, and recurrence.

IPD SHARING:
Plan to Share IPD: No
The medical recoreds were saved in Wan Fang Hospital